CLINICAL TRIAL: NCT01871467
Title: Sargramostim for Myeloid Dendritic Cell Deficiency - Phase I
Brief Title: Sargramostim for Myeloid Dendritic Cell Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KW-5001-1
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Dendritic Cell Deficiency
MeSH Terms: interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sargramostim administration (Experimental): Subjects will receive sargramostim.
  Interventions: Drug: Sargramostim

INTERVENTIONS:
Drug: Sargramostim

SUMMARY:
Previous studies have demonstrated a deficiency of blood dendritic cells in patients with kidney disease that is associated with the development of viral infections after kidney transplantation. We plan to test the ability of sargramostim to increase blood dendritic cell levels in patients with kidney disease in the hopes of developing new therapies to prevent viral infections after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years < 80 years with diagnosis of end stage renal disease and currently undergoing outpatient hemodialysis (HD) at one of the Johns Hopkins University-affiliated HD units

Exclusion Criteria:

* Age<18or>80years
* History of non-adherence to prescribed HD treatment
* Active drug or heavy alcohol use (defined as > 4 drinks/day)
* Pregnancy or breast feeding
* Active infection (bacterial or viral) or clinically significant infections within the past three months (e.g. those requiring hospitalization, or as judged by the PI)
* Active malignancy (with the exception of excised non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin, or adequately treated pre- invasive cervical cancer in situ)
* Unstable cardiovascular status (angina, arrhythmias, congestive heart failure etc...)
* History of liver disease (as defined by a diagnosis of uncompensated cirrhosis) • History of lung disease (including moderate-severe chronic obstructive pulmonary disease, interstitial lung disease, or asthma)
* Known hypersensitivity to yeast-derived products
* Hemoglobin < 10 g/dL and hematocrit < 30%.
* Abnormal white blood cell (WBC) count at baseline (< 3 or > 12 x 10 cells/mm )
* Treatment with WBC growth factors (G-CSF or GM-CSF) or immunosuppressive medications (tacrolimus, cyclosporine, mycophenolate, azathioprine, corticosteroids, chlorambucil, cyclophosphamide) within 4 weeks of study (erythropoiesis-stimulating agents will be allowed)
* Treatment with lithium within 4 weeks of study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Target blood myeloid dendritic cell level of > 2.0 x 10<4>/mL | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl L Womer, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States